CLINICAL TRIAL: NCT06601192
Title: Phase 1, Randomized, Double-Blind Four-Period Crossover, Thorough QT/QTc Study to Evaluate the Effects of EDP-938 on Cardiac Repolarization in Healthy Adults
Brief Title: A Study to Investigate the Effects of Zelicapavir (EDP-938) on QTc Interval in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP 938-008
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: RSV Infection; QTc Interval
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- zelicapavir Dose 1 (therapeutic dose) (Experimental): All participants will receive 4 study interventions. The study interventions will be administered during separate treatment periods starting on Days 1, 9, 17, and 25.
  Interventions: Drug: zelicapavir (therapeutic dose)
- zelicapavir Dose 2 (supratherapeutic dose) (Experimental): All participants will receive 4 study interventions. The study interventions will be administered during separate treatment periods starting on Days 1, 9, 17, and 25.
  Interventions: Drug: zelicapavir (supratherapeutic dose)
- placebo (Placebo Comparator): All participants will receive 4 study interventions. The study interventions will be administered during separate treatment periods starting on Days 1, 9, 17, and 25.
  Interventions: Drug: Placebo
- moxifloxacin (Experimental): All participants will receive 4 study interventions. The study interventions will be administered during separate treatment periods starting on Days 1, 9, 17, and 25.
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: zelicapavir (therapeutic dose) — Subjects will receive zelicapavir (TD) once per treatment period.
  Other Names: EDP-938
  Arms: zelicapavir Dose 1 (therapeutic dose)
Drug: zelicapavir (supratherapeutic dose) — Subjects will receive zelicapavir (SD) once per treatment period.
  Other Names: EDP-938
  Arms: zelicapavir Dose 2 (supratherapeutic dose)
Drug: Placebo — Subjects will receive zelicapavir matching placebo once per treatment period.
  Arms: placebo
Drug: moxifloxacin — Subjects will receive moxifloxin once per treatment period.
  Arms: moxifloxacin

SUMMARY:
The purpose of the study is to assess the effect of a therapeutic and supratherapeutic dose of zelicapavir on the corrected cardiac QT interval relative to a placebo and positive control in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Male or female individuals who are 18 to 65 years of age, inclusive
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Heterosexually active male participants and their female partners of childbearing potential must agree to use 2 effective birth control methods for the duration of the study and for 90 days after the last dose of study intervention.
* Females of childbearing potential must agree to use 2 effective birth control methods for the duration of the study and for 30 days after the last dose of study intervention.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Clinically relevant risk factors for cardiovascular abnormalities
* Pregnant or nursing females
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection
* Infection with HIV, HBV, HCV, or SARS CoV 2
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy)
* Before the first dose of study intervention, participant has received any vaccine, an investigational agent or biological product within 28 days or 5 times the terminal half-life (t½), whichever is longer
* A positive urine drug screen at Screening or Day -1
* Current tobacco smokers or use of tobacco within 3 months prior to Screening
* History of regular alcohol consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Time-matched, placebo-corrected change-from-baseline QTc based on the Fridericia correction QTcF (ΔΔQTcF) after TD and SD of Zelicapavir | Up to 24 hours post dose

SECONDARY OUTCOMES:
Time-matched, placebo-corrected, change-from-baseline non-QT intervals after TD and SD of Zelicapavir | Up to 24 hours post dose
Time-matched, placebo-corrected, change-from-baseline HR after TD and SD of Zelicapavir | Up to 24 hours post dose
Concentration-QTc analysis based on the relationship between plasma concentrations of zelicapavir and ΔΔQTcF after a TD and SD of zelicapavir | Up to 96 hours post dose
Cmax of zelicapavir | Up to 96 hours post dose
Tmax of zelicapavir | Up to 96 hours post dose
t1/2 of zelicapavir | Up to 96 hours post dose
Vd/F of zelicapavir | Up to 96 hours post dose
CL/F of zelicapavir | Up to 96 hours post dose
ΔΔQTcF after moxifloxacin dosing | Up to 24 hours post dose
Safety measured by adverse events | Up to Day 33

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (2):
- United States (2):
  - ICON, Lenexa, Kansas
  - ICON Early Phase, LLC, San Antonio, Texas